CLINICAL TRIAL: NCT01358370
Title: A Retrospective Natural History Study of Patients With Lysosomal Acid Lipase Deficiency/Wolman Phenotype
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LAL-1-NH01
Record Dates: First submitted 2011-04-13; First posted 2011-05-23 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Lysosomal Acid Lipase Deficiency; Wolman Disease
Keywords: LAL Deficiency; LIPA; Wolman disease; Wolman Phenotype; Early Onset LAL Deficiency; Acid Lipase Deficiency
MeSH Terms: conditions — Wolman Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a Natural History study to characterize key aspects of the clinical course of lysosomal acid lipase (LAL) deficiency/Wolman phenotype in patients.

DETAILED DESCRIPTION:
The objective of this study is to characterize key aspects of the clinical course of LAL deficiency/Wolman phenotype in patients including, but not limited to, survival and growth parameters, to serve as a historical control to inform the evaluation and care of affected patients and to provide a reference for efficacy studies of enzyme replacement or other novel therapies.

ELIGIBILITY:
Inclusion Criteria:

* Deceased patients diagnosed with LAL deficiency/Wolman phenotype in 1985 or later provided they have required data points in their medical records.

Exclusion Criteria:

* Patients will be excluded from the study if the required data points for inclusion are not available.
* Living LAL deficiency/Wolman phenotype patients will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Deceased patients diagnosed with LAL deficiency/Wolman phenotype in 1985 or later.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Time to Death | Up to two years.
  The time to death will be analyzed using Kaplan-Meier curves. Estimates (with exact 95% confidence interval [CI]) of the median and the lower and upper quartiles of time to death will be derived.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (7):
  - Cedars-Siani Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - Ney York Presbyterian Hosptial, New York, New York
  - North Shore Long Island Jewish Medical Center, New York, New York
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Hospital Necker- Enfants Malades, Paris, France
- Italy (2):
  - Instituto Giannina Gaslini- Ospedale Pediatrico IRCCS, Genova
  - University of Turin, Turin
- United Kingdom (3):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Kings College London, London
  - Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website — http://alexion.com/